CLINICAL TRIAL: NCT04966806
Title: Contribution of Spherical Aberration and Coma to The Total Ocular High Order Aberration Before and After Femtosecond Laser-Assisted in Situ Keratomileusis Using An Aspheric Ablation Profile
Brief Title: Contribution of SA and Coma to The Total Ocular HOA Before and After FS-LASIK Using An Aspheric Ablation Profile
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Paula Sameh Youssef, Resident., Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PSYoussef
Record Dates: First submitted 2021-06-25; First posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-07

CONDITIONS: FS-LASIK Surgery Effect on Higher Order Aberrations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Percentage of Coma and SA to Total ocular HOA (Other)
  Interventions: Procedure: LASIK refractive surgery

INTERVENTIONS:
Procedure: LASIK refractive surgery — laser vision correction for myopic eyes

SUMMARY:
Laser-assisted in situ keratomileusis (LASIK) is the most frequently performed refractive surgery procedure for the correction of myopia, hyperopia, and astigmatism.

There is a continuous upgrade and development in LVC surgeries correlated with the evolution of new machines and enhancement of the ablation profiles. One of the main undesirable effects of corneal refractive surgeries using conventional ablation profiles is the increase in HOAs which is associated with haloes, glare, ghost images, starburst patterns and monocular diplopia, especially in low lighting conditions and during night driving.

Over the years many ablation profiles have been developed such as wavefront-guided, wavefront optimized, topography guided, Q- Value based and aspheric ablation profiles. These profiles aim to abolish LOAs and to prevent induction or increase of pre-existing HOAs aiming to improve the quality of vision experienced post-operative.

In spite of the vast body of research in this area, there remains a gap in the literature investigating higher-order aberrations' components in-depth. Therefore, this study aims to investigate the contribution of spherical aberration and coma to the total higher order aberration before and after femtosecond assisted laser in situ keratomileusis using an aspheric ablation profile.

This current study is a Descriptive analytical study that was conducted on 34 eyes of 17 patients who underwent corneal refractive surgery.

The results were analyzed to compare the effect of FS-LASIK surgery on corneal coma and SA, and the contribution of each of them on total ocular HOAs preoperative and post-operative.

ELIGIBILITY:
Inclusion Criteria:

1. Age: between 18 years and 45 years
2. Myopes from -1.50 D to -8.00 D
3. Astigmatism less than -4.00 D
4. Normal Corneal Tomography with a Belin Ambrosio big D value of less than 1.6

Exclusion Criteria:

1. Unstable refraction for 1 year
2. Corneal thickness less than 500 microns
3. Expected Post Lasik Residual Stromal bed less than 300 microns
4. All patients with post operative complications as epithelial overgrowth or decentered ablation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2021-07-10 (Estimated); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Change in percentage of contribution of coma and spherical aberration from total ocular HOA before and after FS-LASIK. | 6 months
  Measuring unit for coma and spherical aberrations and total ocular HOA is equivalent Diopters.
  The contribution of coma and spherical aberrations to total ocular HOA will be measured as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al Ainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes